CLINICAL TRIAL: NCT00441051
Title: A Randomized, Double-Blind, Vehicle-Controlled, Single Center, Intra-Individual Comparative Study of the Efficacy and Safety of Diclofenac Sodium 1 mg/g (0.1%) Gel in Subjects With Painful UV-Induced Erythema
Brief Title: Efficacy and Safety of Diclofenac Sodium (0.1%) Gel in Patients With UV Induced Painful Sunburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FESB-DE-310
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Sunburn
Keywords: Sunburn, diclofenac, topical NSAID
MeSH Terms: conditions — Sunburn | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Diclofenac sodium 1mg/g

SUMMARY:
Diclofenac sodium 0.1% will be applied to sunburned skin when the intensity of pain reaches a certain level in order to evaluate the efficacy and safety of the treatment on this induced pain.

ELIGIBILITY:
Inclusion Criteria:

* Have no skin problem which could interfere with the study results or increase the risk of adverse events Have no exposure to excessive or chronic UV radiation (i.e., sunbathing, tanning salon use, phototherapy) within four weeks prior to inclusion, or planned during the study period Have non tanned skin on the areas to be exposed (back) Have a normal tolerance to UV and sun.

Exclusion Criteria:

* Women who are pregnant, planning pregnancy or lactating A known hypersensitivity to diclofenac, aspirin, ibuprofen or other NSAIDs; Use of oral or topical treatments during the month preceding the trial, which may interfere with the results of the trial Other protocol-defined inclusion/exclusion criteria may appl

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2006-11; Study Completion 2006-12

PRIMARY OUTCOMES:
Assess by Visual Analogue Scale (VAS)how products relieve provoked pain (by gloved finger)associated with sunburn in the first 24 hours after UV irradiation.

SECONDARY OUTCOMES:
Assess the spontaneous pain and provoked pain by VAS , the reduction of erythema by erythema scale and chromametry and the safety by reporting adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille- Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Applique a la Dermatologie
Locations (1):
- CPCAD, Nice, France